CLINICAL TRIAL: NCT00179647
Title: A Multicenter, Single-Arm, Open-Label, Expanded Access Program for Lenalidomide With or Without Dexamethasone in Previously Treated Subjects With Multiple Myeloma
Brief Title: Expanded Access Program:Lenalidomide With or Without Dexamethasone In Previously Treated Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Collaborators: Prologue Research International (Industry)
Responsible Party: Robert Knight, MD / Vice President, Clinical Research - Hematology, Celgene Corporation
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-016; NCT00331903 (obsolete NCT alias)
Expanded Access: Available
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2010-03-03 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; MM; Revlimid; CC5013; celgene; cc-5013; relapsed/refractory; lenalidomide; dexamethasone; Decadron
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide 5-25 mg, w/wo dexamethasone (Other): single-arm, open-label, lenalidomide, 5-25 mg, 21/28 days, with/without dexamethasone
  Interventions: Drug: lenalidomide; Drug: dexamethasone

INTERVENTIONS:
Drug: lenalidomide — Lenalidomide, 5 mg to 25 mg, QD, orally, for 21 days every 28 days, with or without dexamethasone
  Other Names: Revlimid
Drug: dexamethasone — Dexamethasone, 20 mg to 40 mg, QD, orally, administered under a variety of dosing regimens
  Other Names: Decadron

SUMMARY:
Subjects who qualify for participation will receive lenalidomide with or without dexamethasone in 4 week cycles until disease progression is documented or lenalidomide becomes commercially available for the indication of multiple myeloma.

DETAILED DESCRIPTION:
This was a multicenter, non-randomized, open-label, uncontrolled, single-arm treatment study of lenalidomide as monotherapy or in combination with dexamethasone in subjects with previously treated relapsed or refractory multiple myeloma, with measurable myeloma paraprotein in serum and/or urine. Subjects who met all of the eligibility criteria were enrolled into the study. Screening procedures took place within 28 days of first dose. Subjects who qualified for participation received oral lenalidomide at a dose of 25 mg daily for 21 days every 28 days.

Subjects had the following options for dexamethasone treatment at the discretion of the treating physician:

Option A: No dexamethasone.

Option B: Oral pulse dexamethasone administered at a dose of 40 mg daily on Days 1-4, 9-12, and 17-20 for each 28-day cycle.

Option C: Oral pulse dexamethasone administered at a dose of 20 mg daily on Days 1-4, 9-12, and 17-20 for each 28-day cycle.

Option D: Oral dexamethasone administered at a dose of 40 mg weekly on Days 1, 8, 15, and 22 for each 28-day cycle for all cycles. Treatment was to be continued as tolerated until disease progression developed.

Doses of lenalidomide were allowed to be reduced first from 25 mg to 15 mg and then in 5-mg decrements due to lenalidomide toxicity. Subjects who could not tolerate a daily dose of 5 mg for 21 days every 28 days were discontinued from treatment. At the discretion of the investigator, doses of dexamethasone were modified due to dexamethasone toxicity. Dose reduction and discontinuation schemes for dexamethasone varied according to the treatment option administered.

Study visits occurred every 2 weeks for the first 3 cycles of therapy and then every 4 weeks after the third cycle until disease progression was documented, study drug was discontinued for another reason, or lenalidomide became commercially available for this indication.

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign an informed consent form.
2. Must be > or = to 18 years of age at the time of signing the informed consent form.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Must be diagnosed with multiple myeloma that is progressing after at least 2 cycles of anti-myeloma treatment or that has relapsed with progressive disease after treatment.
5. Subjects may have been previously treated with thalidomide and/or radiation therapy. In addition, radiation therapy initiated prior to or at baseline (Day 1) may be given concurrently with study therapy, provided that all other eligibility criteria are satisfied.
6. Measurable levels of myeloma paraprotein in serum (>/=0.5 g/dL) or urine (>/=0.2 g excreted in a 24-hour collection sample).
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
8. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study medication.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or lactating females.
3. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) <1,000 cells/mm3 (1.0 x 109/L)
   2. Platelet count <75,000/mm3 (75 x 109/L) for subjects in whom <50% of the bone marrow nucleated cells are plasma cells.
   3. Platelet count <30,000/mm3 (30x109/L) for subjects in whom >/= 50% of bone marrow nucleated cells are plasma cells.
   4. Serum creatinine >2.5 mg/dL (221 mmol/L)
   5. Serum glutamic oxaloacetic transaminase (SGOT, aspartate transaminase [AST]) or serum glutamic pyruvic transaminase (SGPT, alanine transaminase [ALT]) >3.0 x upper limit of normal (ULN)
   6. Serum total bilirubin >2.0 mg/dL (34 mmol/L)
5. Prior history of malignancies other than multiple myeloma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for >/= 1 year.
6. Known hypersensitivity to thalidomide or dexamethasone.
7. Prior history of uncontrollable side effects to dexamethasone therapy.
8. The development of a desquamating rash while taking thalidomide.
9. Use of any standard/experimental anti-myeloma drug therapy within 28 days of the initiation of study drug treatment or use of any experimental non-drug therapy (e.g., donor leukocyte/mononuclear cell infusions) within 56 days of the initiation of study drug treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1913 (Actual)
Dates: Start 2005-09; Primary Completion 2008-12 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (69):
- United States (63):
  - Mayo Clinic, Scottsdale, Arizona
  - Alta Bates Cancer Center, Berkeley, California
  - Scripps Cancer Center, La Jolla, California
  - Cedar Sinai Medical CenterDept of Medicine, Los Angeles, California
  - Kaiser Permanente Medical Group, San Diego, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - University of ColoradoHealth Science Center, Aurora, Colorado
  - Rocky Mountain Cancer Center-Midtown, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Hematology Oncology, PC, Stamford, Connecticut
  - Delaware Clinical & Laboratory Physicians, PA, Newark, Delaware
  - University of Miami Medical School, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Gulf Coast Oncology, St. Petersburg, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - The Palm Beach Cancer Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University Med CtrDivision of Hem/Onc, Chicago, Illinois
  - Rush Cancer Institute, Chicago, Illinois
  - Indiana Univ Cancer Center Bone Marrow Transplantation Program Indiana Cancer Research Institute, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland Medical Center Greenbaum Cancer Ctr, Baltimore, Maryland
  - Center for Cancer And Blood Disorders, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Jackson Oncology Associates, Jackson, Mississippi
  - Siteman Cancer Center, St Louis, Missouri
  - Deaconess Billings Clinic, Billings, Montana
  - Methodist Cancer Center, Omaha, Nebraska
  - Nevada Cancer Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center-Norris Cotton Cancer Center, Lebanon, New Hampshire
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - SUNY Health Science Center - Brooklyn, Brooklyn, New York
  - North Shore Hematology/Oncology Associates, PC, East Setauket, New York
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - NY Presbyterian Hospital/Weill Medical College-Cornell University, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - New York Medical Center, MBCCOP, The Bronx, New York
  - Carolinas Hematology-Oncology Associates, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Dakota Cancer Institute, Fargo, North Dakota
  - Mid Ohio Oncology & Hematology, Inc., Columbus, Ohio
  - Kaiser Permanente Northwest RegionCenter for Health Research, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Charleston Hematology/Oncology P.A., Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Oncology Assoc, Columbia, South Carolina
  - Avera Research Institute, Sioux Falls, South Dakota
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Intermountain Hematology/Oncology, Salt Lake City, Utah
  - Medical College of Virginis, North Hospital, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Gunderson Clinic, La Crosse, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Oncology Alliance, Milwaukee, Wisconsin
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Leukemia/BMT Program of BCDiv of Hem, Vancouver Gen Hosp, Vancouver, British Columbia
  - Dalhousie University Queen Elizabeth II Health Services Centre, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec

REFERENCES:
- [Derived] Reece D, Song KW, Fu T, Roland B, Chang H, Horsman DE, Mansoor A, Chen C, Masih-Khan E, Trieu Y, Bruyere H, Stewart DA, Bahlis NJ. Influence of cytogenetics in patients with relapsed or refractory multiple myeloma treated with lenalidomide plus dexamethasone: adverse effect of deletion 17p13. Blood. 2009 Jul 16;114(3):522-5. doi: 10.1182/blood-2008-12-193458. Epub 2009 Mar 30. PMID 19332768

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide: This was a multicenter, non-randomized, open-label, uncontrolled, single-arm treatment study of lenalidomide as monotherapy or in combination with dexamethasone in subjects with previously treated relapsed or refractory multiple myeloma, with measurable myeloma paraprotein in serum and/or urine. Subjects who met all of the eligibility criteria were enrolled into the study. Screening procedures took place within 28 days of first dose. Subjects who qualified for participation received oral lenalidomide at a dose of 25 mg daily for 21 days every 28 days.
Period: Overall Study
Arm/Group | Lenalidomide
Started | 1913
Completed | 0 (Subjects participated in study until they presented with reason for discontinuation.)
Not Completed | 1913
Not completed — Adverse Event | 294
Not completed — Lack of Efficacy | 478
Not completed — Withdrawal by Subject | 83
Not completed — Lost to Follow-up | 4
Not completed — Death | 94
Not completed — Other | 960

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 1913
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1090
  >=65 years | 823
Age Continuous [Mean (Standard Deviation); unit: years] | 63.4 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 762
  Male | 1151
Region of Enrollment [Number; unit: participants]
  United States | 1183
  Canada | 730

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events Summarized by System Organ Class, Preferred Term, Severity, Seriousness, and Relationship to Treatment.
Description: Data from all subjects who received any study drug were included in the analysis. Adverse events were classified using the Medical Dictionary for Regulatory Activities (MedDRA) classification system. A subject having the same event more than once was counted only once. Adverse events were summarized by worst NCI (National Cancer Institute) CTCAE (Common Terminology Criteria for Adverse Events) VERSION 3.0 grade. Incidence was defined as the number of subjects who experienced an adverse event within their period of participation in this study.
Time Frame: Median time-on-study=18.3 weeks
Reporting Status: Not Posted

2. Primary Outcome: Overall Incidence of Adverse Events
Description: as for outcome 1
Time Frame: Median time-on-study=18.3 weeks
Population: Subjects who received study drug
Measure: Number; unit: Participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 1913
Participants | 1877

ADVERSE EVENTS:
Time Frame: Median time-on-study=18.3 weeks
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 878/1913
Other Adverse Events (participants affected / at risk) | 1877/1913
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=1913)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
ABDOMINAL HAEMATOMA (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 (7)
ABDOMINAL STRANGULATED HERNIA (Gastrointestinal disorders) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 (3)
ACUTE DIVERTICULITIS (Gastrointestinal disorders) | 2 (2)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 3 (3)
AGITATION (Psychiatric disorders) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 68 (75)
ANGINA PECTORIS (Cardiac disorders) | 6 (7)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 7 (8)
ANURIA (Renal and urinary disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 2 (2)
APPENDICITIS (Gastrointestinal disorders) | 1 (1)
APPETITE DECREASED (Metabolism and nutrition disorders) | 2 (2)
ARRHYTHMIA (Cardiac disorders) | 2 (2)
ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12 (12)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 2 (2)
ARTHRITIS INFECTIVE (Infections and infestations) | 1 (1)
ASEPTIC NECROSIS BONE (Musculoskeletal and connective tissue disorders) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ASPERGILLOSIS (Infections and infestations) | 1 (1)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ASTHENIA (General disorders) | 35 (36)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ATAXIA (Nervous system disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 32 (36)
ATRIAL FLUTTER (Cardiac disorders) | 4 (4)
AZOTAEMIA (Renal and urinary disorders) | 2 (3)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 29 (30)
BACTERAEMIA (Infections and infestations) | 10 (10)
BACTERIAL INFECTION (Infections and infestations) | 1 (1)
BACTERIAL SEPSIS (Infections and infestations) | 2 (2)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1)
BLOOD AMYLASE INCREASED (Investigations) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (3)
BLOOD CREATININE INCREASED (Investigations) | 17 (17)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1)
BLOOD HUMAN CHORIONIC GONADOTROPIN INCREASED (Investigations) | 1 (1)
BLOOD UREA INCREASED (Investigations) | 1 (1)
BONE LESION (Musculoskeletal and connective tissue disorders) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 5 (6)
BRADYCARDIA (Cardiac disorders) | 3 (3)
BRAIN OEDEMA (Nervous system disorders) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BRONCHIECTASIS (Infections and infestations) | 1 (1)
BRONCHIOLITIS (Infections and infestations) | 1 (1)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 10 (10)
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 4 (4)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CACHEXIA (Metabolism and nutrition disorders) | 2 (2)
CANDIDA SEPSIS (Infections and infestations) | 1 (1)
CANDIDAL INFECTION (Infections and infestations) | 1 (1)
CARDIAC AMYLOIDOSIS (Cardiac disorders) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 5 (5)
CARDIAC FAILURE (Cardiac disorders) | 2 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 24 (27)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 4 (4)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1)
CATHETER SEPSIS (Infections and infestations) | 1 (1)
CATHETER SITE CELLULITIS (General disorders) | 1 (1)
CATHETER SITE HAEMORRHAGE (General disorders) | 1 (1)
CELLULITIS (Infections and infestations) | 15 (15)
CENTRAL LINE INFECTION (Infections and infestations) | 3 (4)
CEREBRAL HAEMATOMA (Nervous system disorders) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 (2)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 3 (3)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 10 (10)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
CHEST PAIN (General disorders) | 9 (9)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 7 (8)
CHOLANGITIS (Hepatobiliary disorders) | 2 (2)
CHOLECYSTITIS (Hepatobiliary disorders) | 3 (3)
CHOLELITHIASIS (Hepatobiliary disorders) | 2 (2)
CHONDROCALCINOSIS PYROPHOSPHATE (Musculoskeletal and connective tissue disorders) | 2 (2)
CHRONIC OBSTRUCTIVE AIRWAY DISEASE EXACERBATED (Respiratory, thoracic and mediastinal disorders) | 8 (9)
CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Respiratory, thoracic and mediastinal disorders) | 3 (4)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1)
CLOSTRIDIAL INFECTION (Infections and infestations) | 3 (4)
CLOSTRIDIUM COLITIS (Infections and infestations) | 10 (10)
COLITIS (Gastrointestinal disorders) | 3 (3)
COLONIC FISTULA (Gastrointestinal disorders) | 1 (1)
COLONIC PERFORATION (Gastrointestinal disorders) | 1 (1)
COMA (Nervous system disorders) | 1 (1)
COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 2 (2)
CONFUAIONAL STATE (Psychiatric disorders) | 28 (31)
CONSTIPATION (Gastrointestinal disorders) | 5 (5)
CONTUSION (Skin and subcutaneous tissue disorders) | 2 (2)
CONVULSIONS (Nervous system disorders) | 5 (5)
CORONARY ARTERY DISEASE (Cardiac disorders) | 3 (3)
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (5)
DEAFNESS NEUROSENSORY (Ear and labyrinth disorders) | 1 (1)
DEAFNESS UNILATERAL (Ear and labyrinth disorders) | 1 (1)
DEATH (General disorders) | 3 (3)
DEEP VEIN THROMBOSIS (Vascular disorders) | 52 (52)
DEHYDRATION (Metabolism and nutrition disorders) | 41 (48)
DELERIUM (Psychiatric disorders) | 5 (5)
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 3 (3)
DEPRESSION (Psychiatric disorders) | 3 (3)
DERMATITIS BULLOUS (Skin and subcutaneous tissue disorders) | 1 (1)
DERMATITIS MEDICAMENTOSA (Skin and subcutaneous tissue disorders) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 3 (3)
DIABETIC HYPEROSMOLAR NON-KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 18 (18)
DIFFICULTY IN WALKING (General disorders) | 1 (1)
DIPLOPIA (Eye disorders) | 1 (1)
DISORIENTATION (Psychiatric disorders) | 1 (1)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 (1)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 3 (3)
DIVERTICULITIS (Gastrointestinal disorders) | 2 (2)
DIZZINESS (Nervous system disorders) | 3 (3)
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 (1)
DRUG WITHDRAWAL SYNDROME (General disorders) | 1 (1)
DUODENITIS (Gastrointestinal disorders) | 1 (1)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 42 (46)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 (1)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 4 (7)
EMBOLISM (Vascular disorders) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
ENDOCARDITIS INFECTIVE (Infections and infestations) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 1 (1)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 4 (4)
EPIGLOTTITIS (Infections and infestations) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 2 (2)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
EYE INFECTION (Infections and infestations) | 1 (1)
FAECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 7 (7)
FALL (General disorders) | 7 (7)
FATIGUE (General disorders) | 29 (29)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 64 (75)
FEELING COLD (General disorders) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 3 (3)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
FUNGAL INFECTION (Infections and infestations) | 1 (1)
FUNGAL SEPSIS (Infections and infestations) | 1 (1)
GAIT ABNORMAL (General disorders) | 2 (2)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (2)
GANGRENE (Vascular disorders) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1)
GASTROENTERITIS (Gastrointestinal disorders) | 1 (1)
GASTROENTERITIS BACTERIAL (Infections and infestations) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 20 (20)
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL TRACT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
GOUT (Metabolism and nutrition disorders) | 1 (1)
GRAFT VERSUS HOST DISEASE (Immune system disorders) | 1 (1)
GRAM-POSITIVE BACTERIAL INFECTION (Infections and infestations) | 2 (2)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1)
HAEMATOCRIT DECREASED (Investigations) | 1 (1)
HAEMATOMA (Vascular disorders) | 2 (2)
HAEMOGLOBIN DECREASED (Investigations) | 5 (6)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HEART RATE INCREASED (Investigations) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 1 (1)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 1 (1)
HERNIA (General disorders) | 1 (2)
HERPES ZOSTER (Infections and infestations) | 7 (7)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 5 (5)
HOT FLUSHES (Vascular disorders) | 1 (1)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 4 (5)
HYALITIS (Eye disorders) | 1 (1)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 10 (11)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 16 (16)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 19 (19)
HYPERKALEMIA (Metabolism and nutrition disorders) | 8 (8)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERVISCOSITY SYNDROME (Blood and lymphatic system disorders) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 2 (2)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 6 (7)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOKALEMIA (Metabolism and nutrition disorders) | 11 (12)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 8 (9)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 21 (22)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 7 (7)
ILEUS PARALYTIC (Gastrointestinal disorders) | 5 (5)
ILIAC ARTERY STENOSIS (Vascular disorders) | 1 (1)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 (1)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 1 (1)
INFECTION (Infections and infestations) | 19 (19)
INFLUENZA (Gastrointestinal disorders) | 5 (5)
INJECTION SITE THROMBOSIS (General disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 1 (1)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 2 (2)
INTERSTITIAL PNEUMONIA (Infections and infestations) | 1 (1)
INTESTINAL MASS (Gastrointestinal disorders) | 1 (1)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1)
INTRA-ABDOMINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
INTRACTABLE PAIN (General disorders) | 2 (2)
JAUNDICE (Hepatobiliary disorders) | 3 (3)
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 (1)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 (1)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1)
LARGE INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1)
LARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LETHARGY (General disorders) | 4 (4)
LEUKAEMIA PLASMACYTIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 6 (6)
LISTERIOSIS (Infections and infestations) | 3 (3)
LIVER FUNCTION TESTS ABNORMAL (Infections and infestations) | 5 (5)
LOBAR PNEUMONIA (Infections and infestations) | 12 (13)
LOCALISED INFECTION (Infections and infestations) | 5 (6)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4)
LUNG ABSCESS (Infections and infestations) | 1 (1)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LUNG INFECTION (Infections and infestations) | 3 (3)
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 5 (5)
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (2)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MANIA (Psychiatric disorders) | 2 (2)
MEDICATION ERROR (Injury, poisoning and procedural complications) | 5 (6)
MELAENA (Gastrointestinal disorders) | 1 (2)
MENINGITIS (Infections and infestations) | 1 (1)
MENINGITIS PNEUMOCOCCAL (Infections and infestations) | 2 (2)
MENTAL STATUS CHANGES (Psychiatric disorders) | 15 (15)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
METASTASES TO BRAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTASES TO SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
MICTURITION DISORDER (Renal and urinary disorders) | 1 (1)
MIGRAINE WITH AURA (Nervous system disorders) | 1 (1)
MOOD ALTERATION (Psychiatric disorders) | 1 (1)
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
MUCORMYCOSIS (Infections and infestations) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 5 (5)
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 50 (50)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE TWITCHING (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 7 (8)
MYCOBACTERIUM AVIUM COMPLEX INFECTION (Infections and infestations) | 1 (1)
MYELITIS (Nervous system disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 14 (14)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 11 (11)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2)
NECROTISING FASCIITIS (Infections and infestations) | 2 (2)
NEPHRITIS INTERSTITIAL (Renal and urinary disorders) | 1 (1)
NEUROLOGICAL SYMPTOMS (Nervous system disorders) | 1 (1)
NEUROPATHIC PAIN (Nervous system disorders) | 1 (1)
NEUROPATHY (Nervous system disorders) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 45 (46)
NEUTROPENIC SEPSIS (Infections and infestations) | 9 (9)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
OEDEMA (General disorders) | 3 (3)
OEDEMA PERIPHERAL (General disorders) | 2 (2)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1)
OLIGURIA (Renal and urinary disorders) | 1 (1)
OPPORTUNISTIC INFECTION (Infections and infestations) | 2 (2)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1)
ORAL INFECTION (Infections and infestations) | 1 (1)
ORGAN FAILURE (General disorders) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 2 (2)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 5 (5)
OXYGEN SATURATION DECREASED (Investigations) | 2 (2)
PAIN (General disorders) | 14 (16)
PAIN IN LIMB (Musculoskeletal and connective tissue disorders) | 3 (4)
PAIN TRAUMA ACTIVATED (Injury, poisoning and procedural complications) | 1 (1)
PALATAL DISORDER (Gastrointestinal disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 5 (5)
PANCYTOPENIA (Blood and lymphatic system disorders) | 31 (31)
PANIC ATTACK (Psychiatric disorders) | 1 (1)
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 2 (2)
PAROTITIS (Infections and infestations) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 5 (5)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
PEPTIC ULCER (Gastrointestinal disorders) | 1 (1)
PEPTIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 2 (2)
PERFORMANCE STATUS DECREASED (General disorders) | 1 (1)
PERICARDITIS (Cardiac disorders) | 1 (1)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1)
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 (1)
PERIPHERAL NEUROPATHY (Nervous system disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1)
PERIPHERAL SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1)
PERITONSILLAR ABSCESS (Infections and infestations) | 1 (1)
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PLASMACYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 20 (21)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (3)
PNEUMOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1)
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 1 (1)
PNEUMOCYSTIS CARINII PNEUMONIA (Infections and infestations) | 3 (3)
PNEUMONIA (Infections and infestations) | 168 (189)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 5 (5)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1)
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 1 (1)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 2 (2)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 2 (2)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 7 (7)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 6 (6)
POLYDIPSIA (Metabolism and nutrition disorders) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PROTHROMBIN TIME PROLONGED (Investigations) | 1 (1)
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 (1)
PSOAS ABSCESS (Infections and infestations) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 2 (2)
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 29 (29)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PULMONARY OEDEMA (Cardiac disorders) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PYREXIA (General disorders) | 68 (74)
RADIATION OESOPHAGITIS (Injury, poisoning and procedural complications) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 5 (5)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 (1)
RECTAL ABSCESS (Infections and infestations) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3)
RECTOVAGINAL FISTULA (Gastrointestinal disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 31 (32)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 41 (45)
RENAL FAILURE ACUTE ON CHRONIC (Renal and urinary disorders) | 3 (3)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 2 (2)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1)
RENAL MASS (Renal and urinary disorders) | 1 (1)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 2 (2)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 5 (5)
RESPIRATORY DEPRESSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 3 (3)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 13 (13)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (8)
RETINAL VEIN THROMBOSIS (Eye disorders) | 1 (1)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 2 (2)
RIGORS (General disorders) | 7 (7)
RUPTURED DIVERTICULUM (Gastrointestinal disorders) | 1 (1)
SALMONELLA BACTERAEMIA (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 39 (39)
SEPTIC SHOCK (Infections and infestations) | 17 (17)
SICK SINUS SYNDROME (Cardiac disorders) | 3 (3)
SIMPLE PARTIAL SEIZURES (Nervous system disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2)
SINUSITIS (Infections and infestations) | 3 (3)
SINUSITIS ACUTE (Infections and infestations) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE ABSCESS (Infections and infestations) | 1 (1)
SKIN BLEEDING (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 (3)
SOMNOLENCE (Nervous system disorders) | 3 (3)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 6 (6)
SPINAL CORD COMPRESSION (Nervous system disorders) | 12 (12)
SPINAL EPIDURAL HAEMORRHAGE (Nervous system disorders) | 1 (1)
SPONDYLOLISTHESIS ACQUIRED (Musculoskeletal and connective tissue disorders) | 1 (1)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 2 (2)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 2 (2)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 3 (3)
STATUS EPILEPTICUS (Nervous system disorders) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 2 (2)
STREPTOCOCCAL SEPSIS (Infections and infestations) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1)
SUPERIOR VENA CAVAL OCCLUSION (Vascular disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 20 (22)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 2 (2)
TACHYCARDIA (Cardiac disorders) | 2 (2)
THERAPEUTIC AGENT POISONING (Injury, poisoning and procedural complications) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 79 (92)
THROMBOPHLEBITIS (Vascular disorders) | 1 (1)
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 2 (2)
THROMBOSIS (Vascular disorders) | 4 (4)
THROMBOTIC STROKE (Nervous system disorders) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
TONSILLITIS ACUTE (Infections and infestations) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 1 (1)
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 5 (5)
TROPONIN (Investigations) | 1 (1)
TROPONIN INCREASED (Investigations) | 1 (1)
TUMOUR ASSOCIATED FEVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
ULCER (General disorders) | 1 (1)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 10 (10)
URETHRAL HAEMORRHAGE (Renal and urinary disorders) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 2 (2)
URINARY RETENTION (Renal and urinary disorders) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 22 (22)
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 1 (1)
UROSEPSIS (Infections and infestations) | 5 (5)
VASOVAGAL ATTACK (Nervous system disorders) | 2 (2)
VENOUS PRESSURE JUGULAR INCREASED (Investigations) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 (2)
VIRAL INFECTION (Infections and infestations) | 1 (1)
VISUAL DISTURBANCE (Eye disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 16 (16)
WEIGHT DECREASED (Investigations) | 2 (2)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 2 (2)
WOUND INFECTION (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lenalidomide (N=1913)
ANAEMIA (Blood and lymphatic system disorders) | 423 (606)
ANOREXIA (Metabolism and nutrition disorders) | 195 (221)
APPETITE DECREASED (Metabolism and nutrition disorders) | 111 (118)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 218 (267)
ASTHENIA (General disorders) | 277 (338)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 276 (322)
CONFUSIONAL STATE (Psychiatric disorders) | 100 (116)
CONSTIPATION (Gastrointestinal disorders) | 471 (540)
CONTUSION (Skin and subcutaneous tissue disorders) | 123 (154)
COUGH (Respiratory, thoracic and mediastinal disorders) | 301 (349)
DIARRHOEA (Gastrointestinal disorders) | 430 (572)
DIZZINESS (Nervous system disorders) | 261 (321)
DYSGEUSIA (Nervous system disorders) | 171 (185)
DYSPEPSIA (Gastrointestinal disorders) | 129 (148)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 296 (355)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 98 (110)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 114 (129)
FATIGUE (General disorders) | 1072 (1448)
HEADACHE (Nervous system disorders) | 173 (211)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 127 (189)
HYPOAESTHESIA (Nervous system disorders) | 106 (120)
INSOMNIA (Psychiatric disorders) | 386 (424)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 490 (713)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 146 (183)
NASOPHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 161 (209)
NAUSEA (Gastrointestinal disorders) | 362 (455)
NEUROPATHY (Nervous system disorders) | 149 (189)
NEUTROPENIA (Blood and lymphatic system disorders) | 618 (1185)
OEDEMA PERIPHERAL (General disorders) | 285 (371)
PAIN IN LIMB (Musculoskeletal and connective tissue disorders) | 136 (162)
PERIPHERAL NEUROPATHY (Nervous system disorders) | 104 (123)
PYREXIA (General disorders) | 233 (297)
RASH (Skin and subcutaneous tissue disorders) | 273 (368)
STOMATITIS (Gastrointestinal disorders) | 123 (140)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 408 (725)
TREMOR (Nervous system disorders) | 198 (236)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 250 (325)
VISION BLURRED (Eye disorders) | 154 (164)
VOMITING (Gastrointestinal disorders) | 142 (187)
WEIGHT DECREASED (Investigations) | 115 (126)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present the clinical data generated from the study provided that such Investigator shall furnish sponsor with a copy of the proposed publication or presentation at least 60 days in advance of submission, delete any confidential information, and delay submission for up to 90 days to permit the preparation and filing of appropriate intellectual property applications.